CLINICAL TRIAL: NCT05698173
Title: Systemic Lupus Erythematosus and Accelerated Aging
Acronym: LUPAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/53
Record Dates: First submitted 2022-12-21; First posted 2023-01-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Aging
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic Lupus Erythematosus (Experimental): Diagnosis of systemic lupus erythematosus according to American College of Rheumatology (ACR) or SLICC criteria
  Interventions: Biological: blood sample
- Controls (Other): Healthy controls
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 48 ml whole blood for Peripheral blood mononuclear cell (PBMC) and serum isolation
  Arms: Systemic Lupus Erythematosus
Biological: blood sample — blood for Peripheral blood mononuclear cell (PBMC) and serum isolation
  Arms: Controls

SUMMARY:
The study aims at evaluating the phenomena of immune system aging in patients with Systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic systemic autoimmune disease characterized by a breakdown of tolerance against nuclear antigens. Thanks to improvements during the last decades in diagnosis, therapeutics and medical care, the lifespan of SLE patients has remarkably increased. However, standardized mortality ratio are still high in this population, with an increased mortality and morbidity associated with cardiovascular events and infectious events. Interestingly, these conditions are more commonly found during old age in the general population, raising the question of the presence of an acceleration of the aging process in SLE patients.

It has been demonstrated that the aging of the immune system, i.e. immunosenescence, is a key player in the development of many age-related diseases. The acceleration of immunosenescence, as it is observed during chronic viral infections for example, could favor the premature occurrence of clinical manifestations of accelerated aging. The exact contribution of such phenomenon in the context of SLE has, so far, never been explored.

Here, the investigators propose to perform a comprehensive study of the phenomena of immune system aging in patients with SLE in comparison to age-matched healthy controls.

The study will recruit 50 SLE patients followed in Bordeaux University Hospital. Among classical disease activity information, blood samples will be collected at study visit to extensively evaluate immune system aging. Fundamental research will be realized on patients' samples. Patients will be included within their usual follow-up. No extra visit will be needed, and blood samples will be drawn at the same time as those drawn for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* male or female;
* age between 18 and 60 years;
* Lupus patient : diagnosis of systemic lupus erythematosus according to ACR or SLICC criteria;
* being affiliated to health insurance;
* willing to participate and to sign informed consent.

Exclusion Criteria:

* pregnant or breastfeeding women;
* persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Absolute numbers of naïve T lymphocytes | At baseline (Day 0)

SECONDARY OUTCOMES:
Absolute numbers of terminally differentiated T lymphocytes | At baseline (Day 0)
Percentages of terminally differentiated T lymphocytes among total lymphocytes | At baseline (Day 0)
Percentages of senescent lymphocytes among total lymphocytes | At baseline (Day 0)
Telomere length in sorted CD4+ and CD8+ T lymphocytes subsets (naïve and memory) | At baseline (Day 0)
Frequency and phenotype of ELA-specific CD8+ T-cells after 10 days of in vitro priming | At baseline (Day 0)
Number of naïve T lymphocytes newly produced by thymus evaluated by T-cell receptor excision circles (TRECs) measurement | At baseline (Day 0)
Concentrations of senescence-associated secretory phenotype (SASP) markers in patients sera | At baseline (Day 0)
Presence or absence of anti-type I interferons autoantibodies in patients sera | At baseline (Day 0)
Measurement of disease activity according to Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | At baseline (Day 0)
Measurement of disease activity according to British Lupus Assessment Group Index 2004 (BILAG-2004) | At baseline (Day 0)
Quantification of organ damage according to SLICC/ACR Damage Index | At baseline (Day 0)
Levels of anti-double stranded DNA in patients sera | At baseline (Day 0)
Levels of complement components C3 and C4 in patients sera | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Noemie GENSOUS, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Médecine Interne et Immunologie Clinique, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No